CLINICAL TRIAL: NCT03872557
Title: Modulating Glucose Tolerance With Dietary Tyrosine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Judith Korner, Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AAAS2124; R01DK104740 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Glucose Tolerance
Keywords: Glucose tolerance; Tyrosine
MeSH Terms: interventions — Tyrosine; tyrosyltyrosine; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tyrosine (TYR) depletion, then oral TYR (Active Comparator): TYR supplementation: Subjects will be directed to avoid consumption of L-DOPA and TYR enriched foods for 48 hours before oral glucose tolerance test (OGTT). On the evening prior to OGTT, subjects will substitute normal meal and snack for three prepackaged tyrosine-phenylalanine-free liquid meals.
  Visit 2. Placement of intravenous catheter for the collection of serial blood samples and an OGTT with supplementation with oral tyrosine supplement. To supplement the OGTT with Tyrosine, the contents of four (4) L-Tyrosine 500 mg capsule are given 45 minutes before the oral glucose solution is administered. The capsules are to be administered with less than eight ounces of water to minimize dilution of gastric acidity.
  Interventions: Dietary Supplement: Tyrosine (TYR) Supplementation
- TYR depletion, then no oral TYR (No Intervention): Subjects will be directed to avoid consumption of L-DOPA and TYR enriched foods for 48 hours before OGTT. On the evening prior to OGTT, subjects will substitute normal meal and snack for three prepackaged tyrosine-phenylalanine-free liquid meals.
  Subsequent Visit 3. This visit will consist of placement of intravenous catheter for the collection of serial blood samples and an OGTT without supplementation with oral tyrosine supplement.

INTERVENTIONS:
Dietary Supplement: Tyrosine (TYR) Supplementation — L-Tyrosine dietary supplement will be provided as 500 mg capsules and 4 (four) 500 mg capsules are to be given before OGTT. The capsules are formed from animal gelatin, and the contents are formulated with magnesium stearate as a flow agent, but without binders, coatings or colorings and also have no added flavorings, sugars, salt, artificial sweeteners, preservatives or salicylates. The capsules are to be administered with less than eight ounces of water to minimize dilution of gastric acidity.
  Arms: Tyrosine (TYR) depletion, then oral TYR

SUMMARY:
Metabolic or Bariatric surgery is an effective treatment for type 2 diabetes mellitus (T2DM) diabetes associated with obesity. There remain some questions about the biochemical mechanism that drive how these surgeries work to reverse hyperglycemia. In the proposed human studies, the investigators will test the hypothesis that the amino acid tyrosine is a key metabolite in regulating blood sugar levels and that manipulation of the amount tyrosine supplied by nutrition is able to achieve some of the metabolic benefits seen in the early post-surgical period following bariatric surgery. The central hypothesis is that that the tyrosine content of the meal challenge affects post-prandial intestinal and plasma dopamine and levodopa and L-3,4-dihydroxyphenylalanine (L-DOPA) levels, which, in turn, impact β-cell insulin secretion and glucose excursions. The investigators now propose to characterize the possible effects of manipulating dopamine and L-DOPA levels in the gut and plasma on glucose tolerance, insulin secretion, and insulin sensitivity in healthy volunteers with a range of body mass indexes (BMIs).

DETAILED DESCRIPTION:
Several biochemical mechanisms explaining how Roux-en-Y Gastric Bypass (RYGB) provides an effective treatment for obesity associated type 2 diabetes mellitus (T2DM) and improves hyperglycemia independently of weight loss have been proposed. Two are of particular interest; a) the hindgut hypothesis suggesting that nutrient delivery to the distal intestine drives the production of "incretins" which enhance insulin secretion (e.g. glucagon-like peptide-1 (GLP-1)), and b) the foregut hypothesis, positing that foregut bypass reduces the secretion of factors (i.e. anti-incretins) that normally defend against hypoglycemia. The investigators have been actively investigating this topic and have developed a hypothesis based on past studies that they wish to test in a limited human clinical study. In addition, preclinical data suggest that there exists a gut-to-beta cell pathway, responsive to nutritional tyrosine, regulating insulin secretion, and this pathway provides a mechanism for the early postoperative improvements in hyperglycemia observed in RYGB.

ELIGIBILITY:
i. Inclusion Criteria

1. Capable of giving written as well as oral informed consent.
2. A fasting plasma glucose level (FPG) < 126 mg/dL (< 7.0 mmol/L) and an Hb1ac in the 5.7-6.4 % range.
3. BMI in the range of 18-45 kg/m2.
4. Normal Complete blood count (CBC), renal and liver function tests.

ii. Exclusion Criteria:

1. Any diabetes medication within previous three (3) months.
2. Fasting plasma Glucose (FPG) >126 mg/dl or HbA1c > 6.4%
3. Current use (or within 6 months) of antipsychotic, anti-anxiety, or antidepressant medications (e.g. monoamine oxidase (MAO) inhibitors, 5-Hydroxytryptophan (5HT) inhibitors, tricyclic antidepressants, L-DOPA), reserpine, β-2-receptor agonists (e.g., terbutaline), steroids, weight loss medication, anticoagulant medication, over-the-counter nutritional supplements other than standard vitamin and mineral supplements
4. History of Phenylketonuria or other inherited disorders of amino acid metabolism.
5. History of movement disorder such as Parkinson's disease or Huntington's disease
6. Cardiovascular, renal, pulmonary, gastrointestinal, migraines or other medical conditions deemed significant by investigators
7. History of/ or psychiatric illness such as major depression, bipolar disease, anxiety or schizophrenia.
8. History of bariatric surgery with the exception of gastric band if the band has been removed
9. Female of child-bearing age, currently pregnant, breastfeeding or not using a form of birth control.
10. Previous or current use of cocaine, methamphetamine, ecstasy (3-4 methylenedioxymethamphetamine (MDMA))
11. Current daily intake of caffeine >500 mg/day (>4-5 cups of coffee; >10 12-oz cans of soda)
12. Consumption of more than 1 alcoholic drink per day or smoking more than 5 cigarettes/day.
13. Systolic Blood Pressure (SBP) > 150 mmHg; Diastolic Blood Pressure (DBP) > 100 mmHg.
14. Recent history (in the past three months) of more than a 3% gain or loss in body wt.
15. Difficulty in swallowing capsules.
16. Concurrent use of antacids or proton pump inhibitors (e.g.,Prilosec Prevacid, dexilant, Aciphex, Protonix, Nexium, Vimovo, Zegerid)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Whole blood glucose level | Up to 120 minutes from baseline
  Glucose concentration versus time profile following glucose challenge define glucose tolerance
Plasma insulin concentration | Up to 120 minutes from baseline
  Plasma insulin concentration versus time profile following glucose challenge define glucose tolerance
Plasma dopamine concentration | Up to 120 minutes from baseline
  Plasma dopamine concentration versus time profile following glucose challenge may affect glucose tolerance
Plasma L-DOPA concentration | Up to 120 minutes from baseline
  Plasma L-DOPA concentration versus time profile following glucose challenge may affect glucose tolerance
L-tyrosine concentration | Up to 120 minutes from baseline
  Plasma L-tyrosine concentration versus time profile following glucose challenge may affect glucose tolerance
Plasma glucagon concentration | Up to 120 minutes from baseline
  Plasma glucagon concentration versus time profile following glucose challenge impacts glucose tolerance
Plasma GLP-1 concentration | Up to 120 minutes from baseline
  Plasma GLP-1 concentration versus time profile following glucose challenge impacts glucose tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korner J, Cline GW, Slifstein M, Barba P, Rayat GR, Febres G, Leibel RL, Maffei A, Harris PE. A role for foregut tyrosine metabolism in glucose tolerance. Mol Metab. 2019 May;23:37-50. doi: 10.1016/j.molmet.2019.02.008. Epub 2019 Feb 27. PMID 30876866

DOCUMENTS (1):
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT03872557/ICF_000.pdf